CLINICAL TRIAL: NCT00368563
Title: A Capacitance and Transepidermal Water Loss Test to Determine the Ability of Sunscreen to Moisturize Skin
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Loreal USA (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: PEN.1010.02
Record Dates: First submitted 2006-08-23; First posted 2006-08-24 (Estimated); Last update posted 2009-02-11 (Estimated); Status verified 2009-02

CONDITIONS: Dry Skin

INTERVENTIONS:
Drug: Helioblock SX

SUMMARY:
To evaluate the ability of 2 Helioblock SX Cream formulations to moisturize skin using capacitance and transepidermal water loss methodology

ELIGIBILITY:
Inclusion Criteria:

* Healthy,male or female subjects 18 years to 55 years of age, with a minimum Stanfield score at baseline of "2" at the forearm sites intended to be assessed in the study
* Female subjects of childbearing potential using a reliable form of contraception during the course of the study(oral contraceptive pill, intrauterine device, bilateral tubal ligation, abstinence, or other reliable forms at the discretion of the Investigator.) or of non childbearing potential(i.e.,post-menopausal(one year without menstrual period), hysterectomy or bilateral ovariectomy)
* Subjects who have read, understood and signed an informed consent
* Subjects who are willing and capable of cooperating to the extent and degree required by the protocol
* Absence of any visible skin diseases which might be confused with a skin reaction from the test material

Exclusion Criteria:

* Subjects with a condition, or in a situation, which in the Investigator's or Sub-Investigator's opinion, may suggest a significant hazard for the subject, may confound the study results, or may interfere with the subject's participation in the study.
* Subjects with known sensitivities to any of the study preparations or to other skin care products
* Subjects who have participated in a clinical research study, including consumer products studies, within the last 30 days prior to enrollment
* Subjects who are currently receiving medication(prescription or OTC) that in the opinion of the Investigator may interfere with the evaluations made in this study (e.g.vasoactive substances)
* Pregnant or nursing females or women who are planning to get pregnant during the study

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Dates: Start 2006-08; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Oddo, B.S., Principal Investigator — Hill Top Research
Locations (1):
- Hill Top Research, Scottsdale, Arizona, United States